CLINICAL TRIAL: NCT06093152
Title: Video Assisted Study of Salbutamol Response in Viral Wheezing
Acronym: ViVi
Status: Recruiting | Type: Observational
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Terhi Tapiainen, Professor of Pediatrics, Head of Pediatric Infectious Diseases and Emergency Department, University of Oulu
Other Study IDs: 223/2021; FIMEA/2023/003954 (Other: FIMEA)
Record Dates: First submitted 2022-07-05; First posted 2023-10-23 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Wheezing
MeSH Terms: conditions — Respiratory Sounds | interventions — Albuterol

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Before salbutamol: Participants before the administration of salbutamol
- After salbutamol: Participants after the administration of salbutamol
  Interventions: Drug: Salbutamol

INTERVENTIONS:
Drug: Salbutamol — Inhaled salbutamol (SABA, selective beta2-adrenergic receptor agonist) 0,1 mg 4-6 puffs 3-4 times every 20 minutes administered by OptiChamber holding chamber.
  Groups: After salbutamol

SUMMARY:
The study is video assisted cross-over study evaluating the effect of inhaled salbutamol in wheeze in children 6-24 months old.

DETAILED DESCRIPTION:
The object of the study is to evaluate the effect of inhaled salbutamol in wheeze in children 6-24 months old.

In despite of the lack of evidence of salbutamol, it is considered the gold standard in acute wheezing. Placebo-controlled study would be unethical so all participants are treated with salbutamol based on current guidelines. Instead, participants serve as control subjects of their own which is executed by a type video assisted cross-over study.

Participants are filmed before and after the treatment. Afterwards a panel of pediatricians not participating in the treatment of the participants independently evaluates the difficulty of the wheeze. Videos are randomly arranged and members of the panel are blinded to the time point (before/after) of videos.

In addition, collected videos are analyzed using machine vision. Biosignals are collected from the videos and evaluated using algorithms in order to show that machine vision can be utilized to evaluate the difficulty of wheezing. The machine vision analysis is compared to the evaluation of the panel of pediatricians.

ELIGIBILITY:
Inclusion Criteria:

* Wheezing
* Salbutamol-treatment in emergency department prescribed

Exclusion Criteria:

* Need for immediate resuscitation
* Immediate transfer to ICU
* Suspicion of pneumonia based on the auscultation finding
* Suspicion of airway foreign body

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants are 6-24 months old children presenting to the emergency department for wheezing.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in modified RDAI | Within 3 hours of study entry
  RDAI = Respiratory Distress Assessment Instrument, modified to not include auscultation findings. Range 0-18. Higher score indicates more difficult respiratory distress. Evaluated by the blinded panel afterwards using collected videos. Videos collected immediately before and after the intervention.

SECONDARY OUTCOMES:
Change in saturation of peripheral oxygen | Within 3 hours of study entry
  Change in saturation measured immediately before and after the intervention.
Change in auscultation finding | Within 3 hours of study entry
  Evaluated by review of medical records (i.e. based on the findings of the physician treating the patient). Assessed as difficult (wheezing lasting all expiration and possibly inspiration in all 4 lung fields), medium (no inspiratory wheezing, lasting all expiratory OR in all lung 4 fields) of mild (no inspiratory wheezing, wheezing not lasting all expiratory and not in all lung fields). Assessed immediately before and after the intervention.
Change in the difficulty of the respiratory distress | Within 3 hours of study entry
  Subjective evaluation of the respiratory distress based on the appearance of the patient on the video. Range 0-10, higher score indicating more difficult respiratory distress. Assessed by the blinded panel afterwards using videos collected immediately before and after the intervention.
Machine-vision assisted analysis of respiratory status | Within 3 hours of study entry
  Machine vision analysis of the difficulty of wheezing (none - mild - difficult). Assessed using videos collected immediately before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Terhi Tapiainen, Professor, Principal Investigator — University of Oulu
Locations (1):
- Department of Pediatrics, Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No